CLINICAL TRIAL: NCT04618692
Title: Prospective Randomized Single-center Trial Comparing Biliary Anastomosis Using Surgical Loupe Versus Microscope in Living Donor Liver Transplantation
Brief Title: Biliary Anastomosis Using Surgical Loupe Versus Microscope in Living Donor Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, mahmut zenciroğlu, Primary researcher, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Organ transplantation 1
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Liver Failure; Liver Diseases; Liver Cancer; Liver Neoplasms; Liver Dysfunction
Keywords: Liver transplantation; Living donor liver transplantation; Biliary anastomosis
MeSH Terms: conditions — Liver Failure; Liver Diseases; Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: The patients will be randomly allocated in the equal groups.İn group 1 biliary anastomosis will be performed using surgical loupes and İn group 2 biliary anastomosis will be performed using microscope.
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Loupes (Active Comparator): In this group , patients will undergo biliary reconstruction using surgical loupe
  Interventions: Other: Surgical Loupes
- Microscope (Active Comparator): In this group , patients will undergo biliary reconstruction using microscope
  Interventions: Other: Microscope

INTERVENTIONS:
Other: Surgical Loupes — Biliary reconstruction will be performed using surgical loupe
  Arms: Surgical Loupes
Other: Microscope — Biliary reconstruction will be performed using microscope
  Arms: Microscope

SUMMARY:
Comparison of biliary complications in right lobe living donor liver transplantation patients undergoing biliary reconstructions using microscope versus surgical loupes .

DETAILED DESCRIPTION:
Liver transplantation (LT) is the most effective treatment modality in patients with end-stage liver disease and it is also established as a viable treatment option in the field of oncology. Living donor liver transplantation (LDLT) using the right lobe (RL) is a major achievement despite its technical challenges, which has created a significant increase in graft supply. While a secure bile duct anastomosis is one of the basic principles of a successful liver transplant procedure, biliary reconstruction remains the Achilles' heel of LDLT because of the high incidence of posttransplant biliary complications associated with significant recipient morbidity and mortality. Some of these complications are related to technical difficulties due to multiple small biliary orifices, particularly in right lobe grafts. In our center, we have been using microsurgical reconstruction technique for duct-to-duct biliary anastomosis in such grafts. The routine use of this technique has been shown to significantly decrease biliary complications in single-center retrospective studies. However, prospective controlled studies comparing microsurgical and standard biliary reconstruction techniques are lacking. In this study, our objective is to compare posttransplant complications of the two techniques of biliary reconstruction in RL LDLT.

40 patients will be included in the study. They will be randomly allocated in the equal groups.İn group 1 biliary anastomosis will be performed using surgical loupes and İn group 2 biliary anastomosis will be performed using microscope. The patients will be followed for one year after the transplant to compare biliary complications.

ELIGIBILITY:
Inclusion Criteria:

* 1.Primary Adult Living donor liver transplant 2.Right lobe grafts with a single biliary orifice

Exclusion Criteria:

* 1.Bile duct diameter < 3mm 2.Biliary costructions with a hepaticojejunostomy 3.Right lobe grafts with multipl biliary orifice

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Biliary complications after living donor liver transplantation | One year
  Incidence of biliary complications after living donor liver transplantation

SECONDARY OUTCOMES:
Biliary complications | One year
  Types of biliary complications
Biliary related morbidity | One year
  Morbidity
Perioperative mortality | Through study completion, an average of 1 year
  Mortality
Time to biliary complications | One year
  Time to biliary complications

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Yan L, Li B, Zeng Y, Wen T, Zhao J, Wang W, Yang J, Xu M, Ma Y, Chen Z, Liu J, Wu H. Introduction of microsurgical technique to biliary reconstruction in living donor liver transplantation. Transplant Proc. 2007 Jun;39(5):1513-6. doi: 10.1016/j.transproceed.2007.01.091. PMID 17580176
- [Background] Lin TS, Concejero AM, Chen CL, Chiang YC, Wang CC, Wang SH, Liu YW, Yang CH, Yong CC, Jawan B, Cheng YF. Routine microsurgical biliary reconstruction decreases early anastomotic complications in living donor liver transplantation. Liver Transpl. 2009 Dec;15(12):1766-75. doi: 10.1002/lt.21947. PMID 19938121